CLINICAL TRIAL: NCT07328282
Title: Comparative Effects Between ELDOA and Spinal Mobilization With Limb Movement in Lumbar Radiculopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/21
Record Dates: First submitted 2025-12-26; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Lumbar Radiculopathy
Keywords: Lumbar Radiculopathy; lumbar pain
MeSH Terms: conditions — Radiculopathy; Low Back Pain

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ELDOA (Experimental): Group A will recieve standard treatment of ELDOA Strengthening will be divided into following phases
  1. Warm up phase:
  2. Strengthening phase:
  3. Cool down phase:
  Interventions: Procedure: ELDOA
- Spinal mobilization with limb movement (Experimental): Group B will receive Standard treatment of spinal mobilzation and limb movement Strengthening will be divided into following phases
  1. Warm up phase:
  2. Strengthening phase:
  3. Cool down phase:
  Interventions: Procedure: Spinal Mobilization with Limb Movement - SMWLM

INTERVENTIONS:
Procedure: ELDOA — Participants will receive a four-week physiotherapy program with three sessions per week. Each session will heat application followed by supervised stretching and strengthening exercises.
  Participants in Group A will receive ELDOA in addition to standard physiotherapy. Each position will be sustained for at least one minute, with gradual progression to the full posture as flexibility and control improve.
  Arms: ELDOA
Procedure: Spinal Mobilization with Limb Movement - SMWLM — Participants will receive a four-week physiotherapy program with three sessions per week. Each session will heat application followed by supervised stretching and strengthening exercises. Participants in Group B will receive spinal mobilization combined with limb movement along with standard physiotherapy. The technique will be repeated three times.
  Arms: Spinal mobilization with limb movement

SUMMARY:
This study examines the comparative effects of ELDOA and Spinal Mobilization with Leg Movement (SMWLM) on lumbar radiculopathy

DETAILED DESCRIPTION:
Participants were randomly assigned into two groups:

Group A, which performed structured ELDOA exercises targeting spinal decompression and postural alignment Group B, which received SMWLM interventions focusing on spinal mobilization combined with controlled leg movements.

Pain, functional disability, and lumbar range of motion were measured using Visual Analog Scale, Oswestry Disability Index, and bubble inclinometer

ELIGIBILITY:
Inclusion Criteria:

* Age 30 -50 years
* both male and female
* Unilateral lumbar radiculopathy
* Posteriolateral mild disc herniation on MRI
* SLR test positive (30 to 70) degree
* crosed SLR test positive
* Slump test positive
* pain and symptoms disturbution in dermatomal pattern of L4 and L5 Exclusion Criteria
* MRI findings indicating i. Spinal instability ii. Significant neuroforaminal stenosis iii. Structural abnormalities requiring surgical intervention (e.g., large disc herniation )
* Clinical findings indicating:

  i. Absence of severe neurological and severe motor weakness (Manual Muscle Testing grades 0, 1, or 2) ii. Signs of cauda equina lesion (e.g., saddle anesthesia, bowel/bladder dysfunction)
* Diagnosed spinal conditions i. Lumbar spondylolisthesis ii. Lumbar spine fracture iii. Spinal stenosis iv. Spinal tumor v. Ankylosing spondylitis
* History of previous spinal surgery Pregnancy

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Functional Disability | baseline, 2nd and 4th week
  Measured by Oswestry Disability Index, a 10-item questionnaire with six response options per item.
Pain Intensity | baseline, 2nd week, 4th week
  Pain severity will be measured using the Visual Analog Scale ranging from 0 (no pain) to 10 (worst imaginable pain).
Lumbar Range of Motion | baseline, 2nd and 4th week
  Lumbar spine range of motion will be assessed using a bubble inclinometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Punjab Province, Pakistan